CLINICAL TRIAL: NCT01390532
Title: Left Ventricular Dyssynchrony: Rest/Stress 3D Blood-Pool Gated D-SPECT Quantification With a High-Speed Dedicated Cardiac Camera Before CRT
Brief Title: Rest/Stress Quantification Of Left Ventricular Dyssynchrony By 3D Gated Blood Pool D-SPECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre Jean Perrin (Other)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0096; 2010-A00265-34 (Registry Identifier: 2010-A00265-34)
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-07

CONDITIONS: Left Ventricular Dyssynchrony
Keywords: Left Ventricular Dyssynchrony; Gated blood-pool; D-SPECT; Pharmacological stress; NYHA III/IV; LVEF < 35 %; QRS > 120 ms; optimal medical treatment; cardiac resynchronization therapy

INTERVENTIONS:
Device: 3D Blood-Pool Gated SPECT (BPGS) with a new designed cardiac imaging camera (DSPECT, Spectrum Dynamics®, Ceasaria, Israel) — Sequential 5 min Gated blood pool D-SPECT acquisition at rest and during last stage of dobutamine and atropin infusion (>85% PHR).
  Rest and stress left ventricular ejection fraction, phase standard deviation and entropy will be determined using a fully automatic commercial software (QBS, Cedars-Sinai, Los Angeles, CA).

SUMMARY:
Cardiac Resynchronization Therapy (CRT) is an established treatment for patients with advanced heart failure and left ventricular dyssynchrony (LVD). Too many patients do not clinically improve with CRT. New LVD markers other than QRS duration are needed.

Study objective : feasibility assessment of rest and real-time stress 3D Blood-Pool Gated SPECT (BPGS) with a new designed cardiac imaging camera (DSPECT, Spectrum Dynamics®, Ceasaria, Israel) to quantify LVD.

DETAILED DESCRIPTION:
Sequential 5 min Gated blood pool D-SPECT acquisition at rest and during last stage of dobutamine and atropin infusion (>85% PHR).

Rest and stress left ventricular ejection fraction, phase standard deviation and entropy will be determined using a fully automatic commercial software (QBS, Cedars-Sinai, Los Angeles, CA).

ELIGIBILITY:
Inclusion Criteria:

Chronic heart failure with LVEF < 35 %, QRS > 120 ms, NYHA III/IV, optimal medical therapy for more than one month.

* Patient with stable hemodynamic for more than one month,
* More than 18-year old man or woman,
* Patient having given his free, inform and signed consent,
* Patient place setting by the social security system,

Exclusion Criteria:

* Psychiatric disorder
* Any contra-indication to Technetium,
* Any contra-indication to dobutamin or atropin
* Personal or family history of sudden death
* Previous severe ventricular arrhythmia
* Obstructive cardiomyopathy, severe aortic stenosis,
* Pulmonary hypertension,
* History of renal, lung, hepatic, cardiac transplantation,
* Pregnant or breast-feeding Woman,
* Patient who can not conform to the requirements of the protocol,
* Patient included in another medical study,

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Left ventricular phase standard deviation.

SECONDARY OUTCOMES:
Left ventricular entropy
Left ventricle ejection fraction
Quality of life.
6-minutes walking test

CONTACTS AND LOCATIONS:
Overall Officials: Bernard CITRON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de CLERMONT-FERRAND, Clermont-Ferrand, France